CLINICAL TRIAL: NCT03903133
Title: Endothelial Monocyte-activating Polypeptide-II as an Endothelial Dysfunction Marker and Its Relation to the Oxidative Stress in Egyptian Sickle Patients
Brief Title: Endothelial Monocyte-activating Polypeptide-II in Egyptian Sickle Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma Soliman Elsayed Ebeid, MD, Professor of Pediatrics, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AinS HOnc 01
Record Dates: First submitted 2016-09-06; First posted 2019-04-04 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Vitamin E; Antioxidants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vitamin E supplementation (Other): vitamin E supplementation for three months (400-600 mg/day) (400 mg/day in those weighed less than 20 kg and 600 mg/day in those weighed at least 20 kg)
  Interventions: Drug: Vitamin E

INTERVENTIONS:
Drug: Vitamin E — vitamin E supplementation for three months (400-600 mg/day) (400 mg/day in those weighed less than 20 kg and 600 mg/day in those weighed at least 20 kg)
  Other Names: Antioxidant

SUMMARY:
This study objectives to assess the role of endothelial monocyte-activating polypeptide II (EMAP II) as a marker of endothelial dysfunction and disturbed angiogenesis in sickle cell disease and to identify its correlation With the oxidative status.

DETAILED DESCRIPTION:
Study design:

Screening/Baselie Phase

* Detailed medical history with special emphasis on demographic data, transfusion and chelation therapy, disease modifying therapy
* Thorough clinical examination
* Laboratory investigations to be done will include:

  * Liver function test
  * Marker of hemolysis
  * Serum ferritin .
  * Complete blood count(CBC)
  * Hemoglobin electrophoresis
  * Determination of serum levels of EMAP II
  * Lipid Peroxidation (Malondialdehyde Concentration.), Superoxide Dismutase activity, Catalase activity, Glutathione Peroxidase activity, Glutathione Reductase activity, Vitamin E concentration, GSH

The patients under investigations will receive vitamin E supplementation for three months

Patients will be followed up for clinical assessment lying stress on frequency and severity of sickling crisis, length of hospital admission, and frequency and severity of painful crisis

The biochemical investigations, EMAPII and oxidative stress biomarkers will be measured also after the three months vitamin E oral administration.

Statistical analysis Result will be expressed as the mean (+/-) standard deviation (SD). For all tests significance was set at P<0.05. All statistical analysis will be performed using software package SPSS version 17.0 (SPSS Inc,Chicago, IL, USA). Differences over time will be tested with analysis covariance (ANOVA) repeated measures. Repeated measures analysis will be used to test treatment and time effects in addition to group -by- time interaction for clinical laboratory parameters. In cases where interactions will be identified, post hoc comparisons will be adjusted using Bonferroni correlations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell disease as confirmed by qualitative and quantitative analysis of hemoglobin using high performance liquid chromatography (HPLC) at their steady state.

Exclusion Criteria:

* Patients with any inflammatory condition within one month prior to enrollment.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Oxidative stress markers | Two years

SECONDARY OUTCOMES:
Endothelial monocyte-activating polypeptide II | Two year

CONTACTS AND LOCATIONS:
Overall Officials: Fatma SE Ebeid, MD, Principal Investigator — Ain Shams University, Faculty of Medicine

IPD SHARING:
Plan to Share IPD: Yes